CLINICAL TRIAL: NCT06050421
Title: Evaluating the Efficacy of Radically Open Dialectical Behaviour Therapy (RO-DBT) in Patients With Anorexia Nervosa: a Randomized Controlled Clinical Trial
Brief Title: Radically Open Dialectical Behaviour Therapy in Patients With Anorexia Nervosa
Acronym: RODBT-AN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-TDC-2022-123
Record Dates: First submitted 2023-06-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Anorexia Nervosa; Anorexia Nervosa in Remission; Anorexia Nervosa Restricting Type
Keywords: anorexia nervosa, RODBT
MeSH Terms: conditions — Anorexia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as Usual (TAU) (Other): The TAU condition will follow the standard treatment of the EDs Unit of the HSCSP for AN. This treatment consists of visits with a psychiatrist with a frequency decided according to the clinical situation and, in some cases, nursing follow-up and/or relapse prevention group that takes place twice per month
  Interventions: Other: Treatment As Usual
- TAU + Radically Open Dialectical Behaviour Therapy (RO-DBT) (Experimental): 2. TAU + skills of the RO-DBT: In this treatment branch, a RO-DBT skills training therapy will be added to TAU. Treatment and therapists: RO DBT skills training consists of a 30-week intervention program in which a set of skills specifically designed to treat overcontrol are taught on an ongoing basis. The duration of each session is 2 hours. Table X provides an overall summary of each skill training session content. Detailed and extensive information about the treatment can be found elsewhere [24], [34]. Three clinical psychologists and one psychiatrist will conduct the treatment, all of whom have undergone extensive training in RO DBT. A maximum of two therapists will be in charge of each session, and the same two therapists will go throughout each group intervention. The team will be supervised by an approved RO DBT supervisor to improve therapeutic skills and ensure adherence to the protocol.
  Interventions: Behavioral: Radically Open Dialectical Behaviour Therapy (RO-DBT)
- Healty controls (Other): All controls will complete data collection notebook and will undergo the same neuroimaging acquisition. There will not be follow-up for this group.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Radically Open Dialectical Behaviour Therapy (RO-DBT) — RO-DBT is a transdiagnostic intervention specifically designed to treat a spectrum of disorders characterized by excessive overcontrol such as resistant depression, avoidant and obsessive-compulsive personality disorders, mood disorders, anorexia nervosa and autism spectrum disorder.
  Other Names: non
  Arms: TAU + Radically Open Dialectical Behaviour Therapy (RO-DBT)
Other: Treatment As Usual — he TAU condition will follow the standard treatment of the EDs Unit of the HSCSP for AN. This treatment consists of visits with a psychiatrist with a frequency decided according to the clinical situation and, in some cases, nursing follow-up and/or relapse prevention group that takes place twice per month
  Arms: Treatment as Usual (TAU)
Other: No intervention — All controls will complete data collection notebook and will undergo the same neuroimaging acquisition. There will not be follow-up for this group.
  Arms: Healty controls

SUMMARY:
Randomized controlled clinical trial to evaluate the efficacy of "Radically Open Dialectical Behaviour Therapy" in patients with eating disorders: a proof-of-concept study.

DETAILED DESCRIPTION:
Background: Up to 20% of patients with anorexia nervosa (AN) die and 50% relapse after the first episode, being its treatment a great challenge for clinicians. Most therapies excessively focus excessively on nourishment, which translates to temporarily restored weight with no improvements in psychosocial life. Radically Open Dialectical Behaviour Therapy (RO-DBT) is a transdiagnostic treatment designed to treat overcontrol, a key aspect in the functioning of patients with AN. To date no clinical trial (CT) has proved its efficacy on these patients or has demonstrated its biological underpinning mechanisms.

Methods: A randomized CT in AN patients will be conducted, where one group will receive treatment as usual (TAU) and the other one TAU with plus RO-DBT, being psychosocial adjustment the main outcome; other secondary variables will be ED symptoms, overcontrol characteristics, autistic traits and neuroimaging changes.

Discussion: The results will fill the a knowledge gap in AN treatment, expecting that patients who receive TAU with RO-DBT will have better social adjustment and less relapses at one year follow up. This is the first study examining neuroimaging changes in RO-DBT to better understand its underlying mechanisms

ELIGIBILITY:
Inclusion Criteria:

* female patients
* aged between 18 to 65 years old,
* having a diagnosis of AN (DSM 5 criteria),
* having had weigh restoration treatment (normal BMI considered >19 kg/m2)
* having an overcontrol personality style assessed with the styles of coping Word-Pair Checklist scale (ASC-WP)

Exclusion Criteria:

* diagnosis of severe mental illness (schizophrenia or other psychosis, bipolar disorder, major depressive disorder, substance use disorder)
* diagnosis of borderline personality disorder (BPD) or positive result in McLean Screening Instrument for BPD
* mental retardation
* being under standardized psychotherapy at the baseline
* being illiterate or not able to understand Spanish language,
* being left-handed
* being pregnant for MRI requirements.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 90% of people who have AN are women
Enrollment: 96 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire, Q-LES-Q | 6 months
  A self report questionarie that assesses quality of life. The range of scores is 0-100. Higher scores mean higher quality of life.
Quality of Life Enjoyment and Satisfaction Questionnaire, Q-LES-Q | 12 months
  A self report questionarie that assesses quality of life. The range of scores is 0-100. Higher scores mean higher quality of life.

SECONDARY OUTCOMES:
Clinical relapses | 6 months, 12 months
  having BMI below 19kg/m2 during two or more weeks, and having a punctuation of the EAT above 21.
Eating Disorder Inventory, EDI | 6 months, 12 monghs
  A self report questionarie that assesses eating disorder symptomatology. The range of scores is 0-192. Higher scores mean higher eating disorders sympthoms
Autism-Spectrum Quotient, AQ | 6 months, 12 months
  A self report questionarie that assesses autistic traits. The range of scores is 0 to 50. Higher scores mean higher autistic traits.
Rosenberg Self-Esteem Scale, RSE. | 6 months, 12 months
  A self report questionarie that assesses self steem. The scale ranges from 0-30. Higher scores mean higher self-esteem. The range scores is 0-60.
Inventory of Interpersonal Problems (IIP-64) | 6 months, 12 months
  A screening measure for avoidant personality disorder (AVPD), and for personality disorder (PD) in general.
Social Connectedness Scale-Revised, SCS-R | 6 months, 12 months
  This scale assesses the degree to which a person feel connected to others in their social environment. Scores range from 20 to 120 higher score indicates more connectedness to others.
Depression Anxiety and Stress Scale 21 (DASS-21) | 6 months, 12 months
  A self-report scale designed to measure the negative emotional states of depression, anxiety and stress.
Neuroimaging variables | 6 months, 12 months
  structural and functional magnetic resonance images will be acquired at baseline and at 1- month follow-up for all the participants, and in one single occasion for the healthy control group.
Clinical Outcomes in Routine Evaluation-Outcome Measure, CORE-OM, | 6 months, 12 months
  A self-report measure of psychological distress designed to be administered during a course of treatment to determine treatment response. The broad spectrum nature of the measure means it captures a wide variety of problems associated with mental health difficulties, beyond typical symptom measures.
Assessed with the Questionnaire envy in adults, CEA | 6 months, 12 months
  This is composed of 24 items representing all theoretical dimensions. Higher scores show higher envy.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Carmona, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch TR, Gray KL, Hempel RJ, Titley M, Chen EY, O'Mahen HA. Radically open-dialectical behavior therapy for adult anorexia nervosa: feasibility and outcomes from an inpatient program. BMC Psychiatry. 2013 Nov 7;13:293. doi: 10.1186/1471-244X-13-293. PMID 24199611
- [Background] Chen EY, Segal K, Weissman J, Zeffiro TA, Gallop R, Linehan MM, Bohus M, Lynch TR. Adapting dialectical behavior therapy for outpatient adult anorexia nervosa--a pilot study. Int J Eat Disord. 2015 Jan;48(1):123-32. doi: 10.1002/eat.22360. Epub 2014 Oct 27. PMID 25346237
- [Background] Isaksson M, Ghaderi A, Ramklint M, Wolf-Arehult M. Radically open dialectical behavior therapy for anorexia nervosa: A multiple baseline single-case experimental design study across 13 cases. J Behav Ther Exp Psychiatry. 2021 Jun;71:101637. doi: 10.1016/j.jbtep.2021.101637. Epub 2021 Jan 12. PMID 33524917
- [Derived] Avila-Parcet A, Martin-Blanco A, Gawron L, Cano M, Pena-Arteaga V, Carceller-Sindreu M, Soler J, Portella MJ, Faustino G, Cardoner N, Carmona I Farres C. Evaluating the efficacy of radically open dialectical behavior therapy (RO-DBT) in patients with anorexia nervosa: study protocol for a randomized controlled clinical trial. BMC Psychiatry. 2025 Apr 18;25(1):403. doi: 10.1186/s12888-025-06854-9. PMID 40251556